CLINICAL TRIAL: NCT06294639
Title: Median Effective Dose (ED50) of Esketamine Combined With Alfentanil for Children to Inhibit Body Movement During Laser Treatment for Facial Lesion
Brief Title: ED50 of Esketamine for Laser Treatment in Children
Acronym: ESCALATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: XJA-20240224
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia
Keywords: esketamine; children; half effective dose; laser treatment
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Intervention Model Description: The Biased coin method is used
Masking Description: Esketamine will be prepared by an investigator who is not involved in anesthesia and outcome assessment. For all participants, esketamine will be diluted to the same volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- esketamine (Experimental): esketamine will be given intravenously
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — esketamine will be given intravenously
  Other Names: intravenous esketamine

SUMMARY:
There is limited research on the combined use of esketamine and alfentanil for anesthesia during facial laser treatment in pediatric patients, and the effective dosage of esketamine for inhibiting body movement remains unclear. We explore the effective dose of esketamine combined with alfentanil for the inhibition of body movement during facial laser treatment in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* age between 3 years and 12 years old
* patients scheduled for laser treatment of facial lesion

Exclusion Criteria:

* patients with airway infection during the last 1 month
* patients with cardiac or pulmonary disorder
* patients with hepatic or renal disfunction
* patients with neurologic or psychiatric disorder

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-03-27 (Estimated); Primary Completion 2025-03-27 (Estimated); Study Completion 2025-04-27 (Estimated)

PRIMARY OUTCOMES:
half effective dose of inhibition of body movement | from injection of esketamine to start of laser treatment, in an average of 5 minutes

SECONDARY OUTCOMES:
number of patients with agitation during awake | from end of injection of esketamine to 30 minutes after laser treatment, in an average of 60 minutes
number of patients with dizzy during awake | from end of injection of esketamine to 30 minutes after laser treatment, in an average of 60 minutes
number of patients with nausea and vomiting during awake | from end of injection of esketamine to 30 minutes after laser treatment, in an average of 60 minutes
number of patients with apnea during awake | from end of injection of esketamine to 30 minutes after laser treatment, in an average of 60 minutes
satisfaction score of the parents to the anesthesia | from end of laser treatment to discharge from the outpatient unit, in an average of 60 minutes
  The satisfaction of the parents to the anesthesia will be assessed by visual analogue scale, of which 0 is for extremely not satisfied, 10 is for extremely satisfied

IPD SHARING:
Plan to Share IPD: Yes
The data could be shared with request to Prof. Zhihong Lu after publication of the results
Supporting Information: Study Protocol
Time Frame: after publication of the results
Access Criteria: sending email to deerlu23@163.com

REFERENCES:
- [Background] Zhang B, Li M, Han Y, Zhao X, Duan C, Wang J. Effective dose of propofol combined with intravenous esketamine for smooth flexible laryngeal mask airway insertion in two distinct age groups of preschool children. BMC Anesthesiol. 2024 Feb 5;24(1):50. doi: 10.1186/s12871-024-02421-z. PMID 38317070
- [Background] Su M, Zhu Y, Liu S, Song L, Qu J, Zhang Y, Zhang Q. Median effective dose (ED50) of esketamine combined with propofol for children to inhibit response of gastroscope insertion. BMC Anesthesiol. 2023 Jul 18;23(1):240. doi: 10.1186/s12871-023-02204-y. PMID 37464290
- [Background] Zheng XS, Shen Y, Yang YY, He P, Wang YT, Tao YY, Zheng JJ, Sun Y. ED50 and ED95 of propofol combined with different doses of esketamine for children undergoing upper gastrointestinal endoscopy: A prospective dose-finding study using up-and-down sequential allocation method. J Clin Pharm Ther. 2022 Jul;47(7):1002-1009. doi: 10.1111/jcpt.13635. Epub 2022 Mar 7. PMID 35255530